CLINICAL TRIAL: NCT06661811
Title: A Study of CAR-T Cells Targeting B Cell Related Autoimmune Diseases
Brief Title: A Study of CAR-T Cells Targeting Autoimmune Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AID02
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T treatment (Experimental)
  Interventions: Drug: CAR-T

INTERVENTIONS:
Drug: CAR-T — CAR-T cells

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CAR-T cell therapy in patients with autoimmune disease.

DETAILED DESCRIPTION:
Autoimmune disease refers to the disease in which the immune system reacts to the host's own body and causes damage to tissues and organs.

Autoreactive B cells can self-activate and differentiate into plasma cells releasing large amounts of autoantibodies, while they can also present their own antigens to autoimmune T cells, thus activating T cells and promoting the release of inflammatory factors.

CAR-T cells can theoretically completely deplete abnormal antibody-producing B cells, allowing immune rebuilding and restoring the patient's normal immune function, achieving drug-free survival, which fully reflects the application prospects of CAR-T therapy in autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 56 years old;
2. Diagnosed with Autoimmune Diseases；
3. Good organ functions;
4. Voluntary participates this trial and can comprehend and sign ICF.

Exclusion Criteria:

1. Had or has active malignancy;
2. Had been subjected to treatment by CD19 targeted therapy or CAR-T therapy or any gene therapy;
3. Combined with other autoimmune disease that needs treatment;
4. Pregnant or lactating women;
5. Has other factors that deemed not suitable by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2028-04-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 0~28 day after treatment
Frequency of AEs, SAEs | 0 day to 24 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yajing Zhang, MD/PhD, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing Gaobo Boren Hospital, Beijing, China